CLINICAL TRIAL: NCT02336776
Title: Effects of Functional Electrical Stimulation on Muscle Architecture of Patients With Chronic Kidney Disease: Randomized Clinical Trial
Brief Title: Functional Electrical Stimulation in Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FESCKD
Record Dates: First submitted 2015-01-07; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Electrical Stimulation
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional electrical stimulation group (Experimental): Functional electrical stimulation: 80 Hz frequency, 0.4 ms pulse, 10 s time on, 50-20s time off, intensity as patient tolerance, total session time ranged from 20 to 34 minutes.
  Interventions: Other: Functional electrical stimulation
- Control group (No Intervention): The patients in this group were evaluated at baseline and reassessed after eight weeks of follow-up.

INTERVENTIONS:
Other: Functional electrical stimulation — Functional electrical stimulation will be applied through self adhesive electrodes on the quadriceps muscle of both thighs, and these will be positioned at 60° of flexion and contained by a band for that exercise happen isometric form.
  Parameter settings in the electrical stimulator are as follows: 80 Hz frequency, 0.4 ms pulse, 10 s time on, 50-20 s time off, intensity according to the patient's tolerance but enough to cause visible muscle contraction. The total time of each session starts at twenty minutes and is increased every week a total thirty-four minutes at the end of the eighth week. Intervention will be held three times a week for eight weeks and during hemodialysis session.
  Other Names: FES
  Arms: Functional electrical stimulation group

SUMMARY:
Chronic kidney disease is a renal injury and progressive and irreversible loss of kidney function and in its most advanced stage is called chronic renal failure.

Although hemodialysis replace some kidney function, patients suffer some alterations characterized by "uremic syndrome" typically expressed by: motor neuropathy and/or autonomic neuropathy, cardiac or musculoskeletal myopathies, peripheral vascular changes, among others. Thereby, the the adoption of physical exercise should be encouraged. However, it is known that the ability to exercise the subject in hemodialysis is low and keeping in mind the weakness of the muscular system in these individuals, the aim of this study is to assess the effects of functional electrical stimulation (FES) on muscle architecture of patients with chronic kidney disease hemodialysis.

For this the following assessments will be performed before and after stimulation: ultrasonography to assess muscle architecture; six-minute walk test to functional capacity; Kidney Disease and Quality of Life - Short Form questionnaire for quality of life; sit and stand test for resistance of the lower limbs; dynamometric by load cell for muscle strength of the lower limbs; flow-mediated dilatation to endothelial function; blood collection for analysis of inflammatory markers and DNA damage.

The subjects will be randomized into two groups, FESG (functional electrical stimulation group) and CG (control group). The first will receive the FES in the quadriceps muscle of both thighs, for eight weeks, three times a week during hemodialysis session. While the control group only will be evaluated and re-evaluated.

Expected results at the end of the protocol with FES are: increased quadriceps muscle thickness; longest distance covered on the six-minute walk test; improved quality of life; increase in resistance of the lower limbs; increased muscle strength of the lower limbs; improved endothelial function; improved inflammatory status and DNA damage.

DETAILED DESCRIPTION:
The research will be developed in the hemodialysis unit of the Santa Clara hospital of Santa Casa de Misericordia de Porto Alegre.

After the selection of patients for eligibility criteria they will be randomized into functional electrical stimulation group or control group. First all patients will be evaluated, and subsequently the patients in the functional electrical stimulation group will be trained three times per week for eight weeks using an electric current called functional electrical stimulation through the stimulator device NEURODYN II, IBRAMED mark, Amparo, Sao Paulo, Brazil.

The sessions took place in the first hour of dialysis and will last at least 20 and maximum of 34 minutes. The parameters selected in the stimulator will be: 80 Hz frequency, 0.4 ms pulse, 10 s time on, 50-20s time off, intensity as patient tolerance. The patient will be positioned supine, the knees will be at 60° flexion through a foam wedge and ankles restrained by a band to make isometric exercise.

Furthermore, the electrodes used to perform the electrical stimulation will adhesive, disposable and hypoallergenic. These will be placed over the motor points of the quadriceps muscle of both legs in order to make the most effective contraction.

At the end of follow-up, both groups will be further evaluated in order to compare.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease on hemodialysis for more than 3 months;
* Clearance of urea during hemodialysis (Kt/V ≥ 1.2).

Exclusion Criteria:

* Cognitive impairment that prevents conducting evaluations, as well as inability to understand and sign the informed consent form;
* Epidermal lesions at the site of application and/or intolerance stimulator and/or skin sensitivity change;
* Patients with recent sequel of stroke;
* Disabling musculoskeletal disease;
* Uncontrolled hypertension (Systolic blood pressure > 230 mmHg and diastolic blood pressure > 120 mmHg);
* Grade IV heart failure (NYHA) or decompensated;
* Uncontrolled diabetes (blood glucose > 300 mg/dL);
* Unstable angina;
* Fever and/or infectious disease;
* Recent acute myocardial infarction (two months);
* Active smokers; Peripheral vascular disease in the lower limbs as deep vein thrombosis or obliterates thromboangiitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | Eight weeks
  Functional capacity will be assessed by the distance walked in six-minute walk test (6MWT).

SECONDARY OUTCOMES:
Muscle architecture | Eight weeks
  Assessment of muscle architecture will take place with the acquisition of ultrasound images of the medialis and lateralis vastus and rectus femorals through an ultrasound device (Vivid-i, GE, USA). After, the thickness of the muscles will be undertaken in the software ImageJ.
Muscle strength of the lower limbs | Four and eight weeks
  Muscle strength will be evaluated by dynamometry by a load cell.
Endurance of the lower limbs | Four and eight weeks
  The endurance of the lower limbs will be assessed by the number of repetitions performed in sit-and-stand test (STST).
Endothelial function | Eight weeks
  Will be used a high-resolution ultrasound machine (Vivid-i, GE, USA) for evaluation of non-invasive blood endothelial function. Endothelial function will be assessed by flow mediated dilation technique.
Inflammatory profile | Four and eight weeks
  The inflammatory profile will be assessed through blood collection and analysis of biochemical and immunological markers such as interleukin 6, tumor necrosis factor, creatine kinase, lactate and C-reactive protein.
DNA damage | Four and eight weeks
  The damage to DNA is analyzed by electrophoresis single (comet technique), where cells are counted by microscopy.
Quality of Life | Eight weeks
  The quality of life will be assessed by questionnaire Kidney Disease and Quality-of-Life Short-Form (KDQOL-SFTM).

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre